CLINICAL TRIAL: NCT00585715
Title: Evaluation of the Candela 1064nm:Nd:YAG Laser for Skin Tightening
Acronym: IH062905
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Candela Corporation (Industry)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D Associate Professor Departments of Dermatology and Surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20065138; 062905 (Other: University of California, Irvine); UCIaward#062905 (Other Grant/Funding Number: Candela Corporation)
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Localized Lipodystrophy
Keywords: Cellulite; Nd:YAG Laser
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Candela DCD with cooling (Experimental): Laser treatment with Candela DCD cooling which produces a cryogenic fluid that cools the epidermis prior to each laser pulse. Treatment will be conducted on either the left or the right thigh, which will also be randomly determined. The contra-lateral side will not be treated and will serve as a control. The laser system to be used in is Candela GentleYAG, a 1064nm Nd:YAG laser. This arm will receive a coolant during the laser procedure.
  Interventions: Device: 1064 nm Nd:YAG laser
- Candela DCD without Cooling (Active Comparator): Laser treatment without cooling before each laser pulse. Treatment will be conducted on either the left or the right thigh, which will also be randomly determined. The contra-lateral side will not be treated and will serve as a control. The laser system to be used in is Candela GentleYAG, a 1064nm Nd:YAG laser. This arm will not receive a coolant during the laser procedure.
  Interventions: Device: 1064 nm Nd:YAG laser

INTERVENTIONS:
Device: 1064 nm Nd:YAG laser — 3 treatments at 3-5 week intervals Spot size: 10 - 18 mm diameter Fluence: 50 J/cm2 Laser pulse duration: 50 ms Rep. rate: Up to 2 Hz DCD cooling 0-50 ms
  Other Names: Candela Gentle YAG Laser

SUMMARY:
The purpose of this research study is to evaluate effectiveness of a non-ablative (does not remove skin) treatment for cellulite (dimpled fat) in conjunction with skin tightening using the Candela GentleYAG laser.

DETAILED DESCRIPTION:
The objective of this investigation is to evaluate the effectiveness of a non-ablative treatment for skin laxity by increasing dermatofibrosis of the reticular dermis using the Candela GentleYAG laser. Treatment areas will be limited to the thighs.

* The primary objective is to assess the safety and efficacy of the laser for improvement in appearance of cellulite.
* The secondary objective is to assess the safety and efficacy of the laser with cooling and the laser without cooling for improvement in appearance of cellulite.

This is an open label trial. Treatment will be conducted on either the left or the right thigh, which will be randomly determined. The contra-lateral side will not be treated and will serve as a control. A comparison of baseline photographs (prior to treatments) to photographs taken 1 and 3 months after the completion of treatments will be conducted. Photographic equipment and the protocol for photography will be consistent at each visit. Ultrasound may be taken at baseline and at the follow-up visits to evaluate flatness of cellulite and dermal fibrosis or enlargement of the reticular dermis. The circumference of the area to be treated will be measured with a tape measure, weight/height will be recorded and the Body Mass Index (BMI) will be calculated at baseline and follow-up visits. In addition, skin elasticity may be measured at the treatment areas at baseline and follow-up visits. The photographs, ultrasound and measurements will be taken using consistent procedures at each visit by viewing the baseline photograph and using landmarks such as freckles and birthmarks.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals, male or female, greater than 40 years of age.
2. Moderate skin laxity in the arms, legs, abdomen, or neck.
3. Subject is not overweight. Body Mass Index (B.M.I.) is ≤ 27.
4. Subject has Fitzpatrick skin phototype I-IV.
5. Subject is willing to participate in study and adhere to follow-up schedule.
6. Subject is able to read and comprehend English.
7. Subject has completed Informed Consent Form.

Exclusion Criteria:

1. Subjects that have had liposuction or other surgical procedures (including mesotherapy) to remove fat in the treatment area during the past year.
2. Subject is overweight (BMI > 27).
3. Subject has known photosensitivity or history of ingesting medications known to induce photosensitivity in the previous 3 months.
4. Subject has a personal or family history of keloid formation or scarring.
5. Subject is pregnant or lactating.
6. Subject has a history of uncontrolled diabetes and/or requires medication which may interfere with the study.
7. Subjects with a known history of neuropathy.
8. Subjects with a known history of a coagulopathy.
9. Subject is unable or unwilling to comply with the study requirements
10. Subject has pacemaker or metallic implants.
11. Subject has Fitzpatrick skin type V and VI.
12. Subject is mentally incompetent or a prisoner.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Kelly, M.D., Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Beckman Laser Institute, Irvine, California
  - UC Irvine Dermatology Clinical Research Center, Irvine, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Truitt, A., Echague, A., Zachary, C. Kelly K.M. Evaluation of the Candela 1064 nm Nd:YAG Laser for Cellulite and Skin Tightening. Presented at the American Society for Laser Medicine and Surgery Annual Meeting, 2007, Dallas, TX.
- See also: UC Irvine Department of Dermatology Clinical Research — http://www.dermatology.uci.edu/clinical_research.html
- See also: Beckman Laser Institute — http://www.bli.uci.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser With Cooling: Laser used with Candela DCD cooling which produces spray of cryogenic fluid that cools the epidermis prior to each laser pulse. Pulse duration 20-50ms using wavelength 1064nm. Laser treatments repeated every 3 weeks for a total of 3 treatments.
- Laser Without Cooling: Laser used without Candela DCD cooling. Pulse duration 20-50ms using wavelength 1064nm. Laser treatments repeated every 3 weeks for a total of 3 treatments.
Period: Overall Study
Arm/Group | Laser With Cooling | Laser Without Cooling
Started | 11 | 11
Completed | 8 | 11
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser With Cooling | Laser Without Cooling | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (9.47724547) | 36 (8.40346249) | 37 (8.77225062)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mild to Moderate Reduction in Cellulite.
Description: Nurnberger-Muller Scale :
  Stage 0: No dimpling. Stage 1: No dimpling. Stage 2: Dimpling spontaneously standing. Stage 3: Dimpling spontaneously standing and lying down.
  Texture Scale:
  Hard or Solid: Pinch test "firm folds and furrows." Adherent to deep planes. Not modified with lying versus standing position.
  Soft or Flaccid: Pinch test "spongy and floating folds and furrows." No adherence to deep planes. Not painful, flaccid. "Orange peel skin" appears spontaneously.
  Edematous: Doughy consistency. Pain and cramps. Signs of venous and lymphatic insufficiency "legs in boot/column".
  At the 6month follow-up, a blinded assessor ranked changes in cellulite appearance on subject's thighs according to the prior cellulite dimpling and texture criteria. Change in cellulite appearance was assessed on a scale of 0-3, with 0 as "no change" and 3 as "significant change." Improvement in cellulite appearance was characterized by an increase of one unit or more on this scale.
Time Frame: 6 month follow up
Population: Only subjects who completed the 6 month follow-up were included in the analysis
Measure: Number; unit: participants
Groups:
- Laser With Cooling for Skin Tightening: Laser used with Candela DCD cooling which produces spray of cryogenic fluid that cools the epidermis prior to each laser pulse. Pulse duration 20-50ms using wavelength 1064nm. Laser treatments repeated every 3 weeks for a total of 3 treatments.
- Laser Without Cooling for Skin Tightening: Laser used without Candela DCD cooling. Pulse duration 20-50ms using wavelength 1064nm. Laser treatments repeated every 3 weeks for a total of 3 treatments.
Arm/Group | Laser With Cooling for Skin Tightening | Laser Without Cooling for Skin Tightening
Number analyzed (Participants) | 7 | 9
participants | 3 | 2

2. Primary Outcome: Average Extent of Reduction in Cellulite Appearance for Patients With Reported Mild to Moderate Cellulite Reduction.
Description: At the 6 month follow-up, a blinded assessor ranked change in cellulite appearance on subject's thighs according to the prior cellulite dimpling and texture criteria. Change in cellulite appearance was assessed on a scale of 0-3, with 0 as "no change" and 3 as "significant change."
  Using this scale, the average reduction in cellulite appearance was calculated for each participant that experienced a mild to moderate reduction in cellulite appearance.
Time Frame: 6 month follow up
Population: The average amount of cellulite reduction was calculated from the 5 subjects who experienced mild to moderate improvement in cellulite appearance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laser With Cooling for Skin Tightening | Laser Without Cooling for Skin Tightening
Number analyzed (Participants) | 3 | 2
units on a scale | 1 (0) | 2 (0)

ADVERSE EVENTS:
Description: There were no adverse events reported.
Arm/Group | Laser With Cooling | Laser Without Cooling
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2009-05-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT00585715/Prot_000.pdf